CLINICAL TRIAL: NCT01381627
Title: Safety Evaluation of Dexmedetomidine Monitored Anesthesia Care for Endobronchial Ultrasound-guided Transbronchial Needle Aspiration
Brief Title: Safety Evaluation of Dexmedetomidine for EBUS-TBNA
Acronym: EBUSed
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Louis-Philippe Fortier, MD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11021
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2011-06

CONDITIONS: Lung Cancer
Keywords: EBUS-TBNA; Dexmedetomidine; Precedex; Remifentanil; Ultiva; Monitored Anesthesia Care; Sedation; Bronchoscopy; Lung cancer; Mediastinal node; Cancer staging; Anesthesia; Remote location
MeSH Terms: conditions — Lung Neoplasms | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Remifentanil IV bolus 0.5 mcg/kg bolus in 10 minutes. Initial bolus followed by infusion 0.05-0.25 mcg/kg/min for OAA/S 2-3. Remifentanil IV bolus 0.3 mcg/kg PRN for time-limited painful stimuli.
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Dexmedetomidine — Dexmedetomidine 0.4 mcg/kg IV bolus in 10 minutes. Dexmedetomidine 0.5-1.0 mcgg/kg/h for OAA/S 2-3. Midazolam 0.015 mg/kg bolus IV PRN.
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
Lung cancer is the second most commonly diagnosed primary neoplasia in Canada accounting for 22 865 new cases in 2007. Recent randomized trials have shown a significantly better diagnostic yield and fewer unnecessary thoracotomies with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) when compared to conventional TBNA for various clinical conditions including peripheral pulmonary lesions and sarcoidosis. EBUS-TBNA are now routinely performed in our institution for staging of pulmonary and mediastinal cancer. EBUS-TBNA are performed under monitored anesthesia care (MAC) in the endoscopy suite at the Centre de soins ambulatoires of the Hôpital Maisonneuve-Rosemont.

Remifentanil, used in combined regime or as single agent proved to be effective and safe for MAC. Nonetheless, anesthesiologists are still confronted to the respiratory depression profile of remifentanil and other commonly used agents. An analysis of the ASA Closed Claims demonstrated that respiratory depression remains a significant drawback during MAC in remote locations. Furthermore, patients with coexisting pulmonary diseases scheduled for EBUS-TBNA are at increased risk of such complications.

The investigators hypothesize that compared to the use of remifentanil-based MAC protocol, the use of dexmedetomidine-based MAC protocol for EBUS-TBNA will result in a lower incidence of major respiratory and hemodynamic adverse events (bradypnea, apnea, oxygen desaturation, hypotension, hypertension, bradycardia and tachycardia) with equivalent overall procedure conditions.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Subjects with planned EBUS-TBNA under conscious sedation.
* Age 18-75 years old.
* American Society of Anesthesiologists class I-III.
* The subject is able to understand the study objectives, the experimental protocol and procedures, and is capable of providing an informed consent.

Exclusion Criteria:

* Subjects allergic to any of the study drugs.
* BMI > 34 kg/m2.
* Severe renal or hepatic failure.
* Pregnancy.
* Emergent procedure.
* Heart failure NYHA > III.
* Systolic blood pressure < 90 mmHg.
* Advanced heart block (unless patient has a pacemaker).
* Unstable angina and/or myocardial infarction within past 6 weeks.
* FEV1 ≤ 0.8 L.
* Oxygen-dependent patient.
* Use of α2-adrenoreceptor agonist or antagonist within 14 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Bradypnea,apnea, oxygen desaturation, hypotension, hypertension, heart rate <45 beats per minute, heart rate ≥120 beats per minute

SECONDARY OUTCOMES:
Vocal cord movement | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Vocal cord movement before fiberscope passage
Sedation scores | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Observer's Assessment of Alertness/Sedation Scale (OAA/S) throughout the EBUS-TBNA procedure. Specific time points: before fiberscope nasal insertion, before vocal cord passage, after vocal cord passage and at the end of the procedure.
Aldrete scores in the post anesthesia care unit | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Aldrete score immediately after removal of fiberscope, time for Aldrete score equal or superior to 9 (assesed at 5 minute intervals).
Nausea and vomiting | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
Cumulative dose of remifentanil or dexmedetomidine | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
Total dose of lidocaine | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Cumulative dose of lidocaine administered by the endoscopist
Total dose of vasopressor | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Cumulative dose of vasopressor administered
Coughing episodes | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Coughing episodes throughout the EBUS-TBNA procedure
Endoscopist satisfaction | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Endoscopist global satisfaction score based on a 4-point Likert scale
Recall | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Recall evaluation once Aldrete score superior to 9 in post anesthesia care unit. Evaluation based on a 4-point Likert scale
Pain associated with the procedure (VAS) | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Maximal pain evaluation based on a visual analog scale. Score measured once an Aldrete score superior to 9 in the post anesthesia care unit is achieved.
Patient satisfaction | Patient followed for the entire duration of EBUS-TBNA (avg. 40 min) and until discharge of PACU (1 day total, ambulatory basis)
  Global patient satisfaction associated with the procedure. Score based on a 5 point Likert scale. Measured before patient leaves the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Verdonck, MD, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Derived] St-Pierre P, Tanoubi I, Verdonck O, Fortier LP, Richebe P, Cote I, Loubert C, Drolet P. Dexmedetomidine Versus Remifentanil for Monitored Anesthesia Care During Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration: A Randomized Controlled Trial. Anesth Analg. 2019 Jan;128(1):98-106. doi: 10.1213/ANE.0000000000003633. PMID 29958220